CLINICAL TRIAL: NCT00718328
Title: Simvastatin For Intracerebral Hemorrhage Study
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Poor recruitment, trial terminated
Sponsor: Johns Hopkins University (Other)
Collaborators: National Center for Research Resources (NCRR) (NIH); National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NA_00016284; NIH UL1 RR 025005
Record Dates: First submitted 2008-07-15; First posted 2008-07-18 (Estimated); Results first posted 2017-06-12 (Actual); Last update posted 2017-10-09 (Actual); Status verified 2017-09

CONDITIONS: Intracerebral Hemorrhage
Keywords: Intracerebral; Hemorrhage; Edema; Statins
MeSH Terms: conditions — Cerebral Hemorrhage; Hemorrhage; Edema | interventions — Simvastatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- I (Experimental): Simvastatin Group
  Interventions: Drug: Simvastatin 80 mg
- II (Placebo Comparator): Placebo Group
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Simvastatin 80 mg — Patients in study arm 1 will receive simvastatin 80 mg once daily for 14 days or until death or discharge.
  Arms: I
Drug: Placebo — Patients in study arm II will receive placebo once daily for 14 days or until death or discharge.
  Arms: II

SUMMARY:
Study Objective: To analyze if statins are effective in ameliorating perihematomal edema evolution thereby reducing mortality and improving functional outcomes following spontaneous intracerebral hemorrhage (ICH).

DETAILED DESCRIPTION:
Intracerebral hemorrhage (ICH) causes 10% to 15% of first-ever strokes, with a 30-day mortality rate of 35% to 52% with only 20% expected to be functionally independent at 6 months. No medical or surgical interventions have been found to alter the natural evolution of this disease. The high risk for mortality and poor outcomes seems to occur despite relatively small hematoma volumes and small amounts of neuronal tissue at risk for injury. The reasons for this observation remain unknown; however perihematomal edema formation and inflammation that follows ICH seems to play an important role.

The Simvastatin for Intracerebral Hemorrhage Study is a prospective double blinded placebo controlled randomized (1:1) clinical trial that compares outcomes in patients receiving generic simvastatin 80 mg for 14 days or until death or discharge with patients in the placebo group.

The hypothesis for our study is that statins ameliorate perihematomal edema evolution thereby reducing mortality and improving functional outcomes following Intracerebral Hemorrhage (ICH). This hypothesis in turn is based on animal data showing suppression of inflammatory reaction and improved neurological outcomes following administration of statins to rodents with experimental ICH, and on a retrospective review of patients admitted to The Johns Hopkins Hospital over the last 7 years with spontaneous ICH which showed significantly better outcomes (decreased 30 day mortality secondary to decreased perihematomal edema) in patients on statins at the time of admission.

ELIGIBILITY:
Inclusion Criteria:

* Patient with CT evidence of ICH admitted within 24 hours of onset of symptoms.

Exclusion Criteria:

* Age < 18 or > 85
* Admission Glasgow Coma Score (GCS) < 6
* ICH volume < 10 cc
* ICH secondary to trauma, aneurysm, Arterio-Venous Malformation (AVM), tumor or post surgical
* Multiple ICH
* Associated Subdural hematoma or significant Subarachnoid hemorrhage
* History of prior neurologic disease with modified Rankin Scale (mRS) > 1
* Hematoma evacuation, hemicraniectomy, clot lysis
* Myopathy
* Active Liver disease
* Pregnancy
* Statin allergy
* Patients on statins prior to admission
* Patients with an acute indication for statin therapy (Unstable angina)

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2008-10; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Neeraj S Naval, M.D., Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Bayview Medical Center, Baltimore, Maryland, United States

REFERENCES:
- [Background] Naval NS, Abdelhak TA, Zeballos P, Urrunaga N, Mirski MA, Carhuapoma JR. Prior statin use reduces mortality in intracerebral hemorrhage. Neurocrit Care. 2008;8(1):6-12. doi: 10.1007/s12028-007-0080-2. PMID 17701108
- [Background] Naval NS, Abdelhak TA, Urrunaga N, Zeballos P, Mirski MA, Carhuapoma JR. An association of prior statin use with decreased perihematomal edema. Neurocrit Care. 2008;8(1):13-8. doi: 10.1007/s12028-007-0081-1. PMID 17701107

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period October 2008- June 2009, Inpatient (ICU)
Pre-assignment Details: No issues prior to assignment
Groups:
- Simvastatin Group: Simvastatin 80 mg: Patients in study arm 1 will receive simvastatin 80 mg once daily for 14 days or until death or discharge.
- Placebo Group: Placebo: Patients in study arm II will receive placebo once daily for 14 days or until death or discharge.
Period: Overall Study
Arm/Group | Simvastatin Group | Placebo Group
Started | 1 | 0
Completed | 0 (Prematurely terminated due to poor enrollment) | 0 (Terminated due to poor enrollment)
Not Completed | 1 | 0
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Simvastatin Group | Placebo Group | Total
Number analyzed (Participants) | 1 | 0 | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 0 | 1
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: years] | 62 [62 to 62] |  | 62 [62 to 62]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 |  | 0
  Male | 1 |  | 1
Region of Enrollment [Number; unit: participants]
  United States | 1 |  | 1

OUTCOME MEASURES:

1. Primary Outcome: Perihematomal Edema
Description: Solitary patient lost to follow up (out of state)
Time Frame: Days 7 and 14
Measure: Mean (Standard Deviation); unit: Relative perihematomal edema
Arm/Group | Simvastatin Group | Placebo Group
Number analyzed (Participants) | 1 | 0
Relative perihematomal edema | NA (NA) — Patient lost to follow up |

ADVERSE EVENTS:
Arm/Group | Simvastatin Group | Placebo Group
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/0
Other Adverse Events (participants affected / at risk) | 0/1 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No